CLINICAL TRIAL: NCT00445211
Title: Heparin Requirement in Counterpulsation
Brief Title: HEROIC (Heparin Requirement in Counterpulsation)
Acronym: HEROIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Justin Trivax, MD Cardiologist, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-001
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Cardiogenic Shock
Keywords: Intraaortic balloon pumping; Heparin; Limb ischemia; Bleeding
MeSH Terms: conditions — Shock, Cardiogenic; Hemorrhage | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intra-Aortic balloon Pump with Heparin (Active Comparator): Intra-Aortic Balloon Pump (IABP) with Heparin
  Interventions: Drug: Heparin
- Intra-Aortic balloon Pump without Heparin (Active Comparator): Intra-Aortic balloon Pump (IABP) without Heparin
  Interventions: Other: Without Heparin

INTERVENTIONS:
Drug: Heparin — Heparin administered at 500units/hour while on Intra-Aortic balloon Pump (IABP).
  Arms: Intra-Aortic balloon Pump with Heparin
Other: Without Heparin — Intra-Aortic balloon Pump (IABP) without Heparin.
  Arms: Intra-Aortic balloon Pump without Heparin

SUMMARY:
Patients with intra-aortic balloon pumps (catheters placed in the groin connected to a pump which assists the heart by opening and closing a balloon in the aorta, thereby decreasing the work of the heart and improving blood flow to the coronary arteries) often receive intravenous (IV) heparin (a "blood thinner") to prevent circulation problems in the leg (where they are inserted). When intra-aortic balloon pumps were initially developed, the catheters were larger than the catheters used today. Due to the large size of the catheter and the material used to make the catheter, it was thought that intravenous heparin would prevent poor blood flow to the leg that contained the temporary catheter. Intravenous heparin, however, has never been proven to maintain good blood flow in these patients. The catheters used with intra-aortic balloon pumps are now smaller in size and made of a material that is less likely to produce blood clots. It is not clear that heparin is needed with intra-aortic balloon pumps. Bleeding complications associated with intra-aortic balloon pumps may be decreased if heparin is not used. In 2004, 99 patients received intra-aortic balloon pumps in the cardiac catheterization labs at William Beaumont Hospital. These patients received intravenous heparin and experienced a large number of bleeding complications (27 patients required a blood transfusion). This study will help the investigators to clarify if heparin should or should not be routinely used in patients with intra-aortic balloon pumps.

DETAILED DESCRIPTION:
Potential patients will be identified in the cardiac catheterization lab when an intra-aortic balloon pump is placed. Patients who agree to participate in this study will be randomized (they will be selected to receive heparin or not to receive heparin with their intra-aortic balloon pump) by a process that is similar to flipping a coin. Patients will have a 50% chance of receiving heparin and a 50% chance of not receiving heparin. If a patient does not want to participate in the study, his/her cardiologist will decide if the patient will receive or not receive heparin. Intra-aortic balloon pumps have been used with and without intravenous heparin and there is no known increase in complications in patients who do not receive heparin. Risks include bleeding and possible blood clots/decreased blood flow to the leg with the catheter in both groups (due to different medical reasons). The patients in both groups will be monitored closely in the cardiac care unit while the intra-aortic balloon pump is in place to prevent and/or minimize complications.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Able to provide consent
* Insertion of Intra-aortic Balloon Pump (IABP) in William Beaumont Hospital (WBH) cath lab
* Anticipated duration of IABP >/= 18 hours

Exclusion Criteria:

* Contraindications to heparin
* Pre-existing condition requiring heparin administration (other than IABP)
* IABP placed outside of the WBH cardiac catheterization lab prophylactically for high-risk percutaneous coronary intervention (PCI), without complications)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Trivax, M.D., Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baim DS, Grossman W. Grossman's Cardiac Catheterization, Angiography and Intervention (6th Ed). Lippincott Williams & Williams, Philadelphia, Pennsylvania, 2000, 463.
- [Background] MOULOPOULOS SD, TOPAZ S, KOLFF WJ. Diastolic balloon pumping (with carbon dioxide) in the aorta--a mechanical assistance to the failing circulation. Am Heart J. 1962 May;63:669-75. doi: 10.1016/0002-8703(62)90012-1. No abstract available. PMID 14476645
- [Background] Kantrowitz A. Origins of intraaortic balloon pumping. Ann Thorac Surg. 1990 Oct;50(4):672-4. doi: 10.1016/0003-4975(90)90220-z. PMID 2222066
- [Background] Stone GW, Ohman EM, Miller MF, Joseph DL, Christenson JT, Cohen M, Urban PM, Reddy RC, Freedman RJ, Staman KL, Ferguson JJ 3rd. Contemporary utilization and outcomes of intra-aortic balloon counterpulsation in acute myocardial infarction: the benchmark registry. J Am Coll Cardiol. 2003 Jun 4;41(11):1940-5. doi: 10.1016/s0735-1097(03)00400-5. PMID 12798561
- [Background] Cohen M, Dawson MS, Kopistansky C, McBride R. Sex and other predictors of intra-aortic balloon counterpulsation-related complications: prospective study of 1119 consecutive patients. Am Heart J. 2000 Feb;139(2 Pt 1):282-7. doi: 10.1067/mhj.2000.101489. PMID 10650301
- [Background] Alle KM, White GH, Harris JP, May J, Baird D. Iatrogenic vascular trauma associated with intra-aortic balloon pumping: identification of risk factors. Am Surg. 1993 Dec;59(12):813-7. PMID 8256934
- [Background] Walls JT, Boley TM, Curtis JJ, Silver D. Heparin induced thrombocytopenia in patients undergoing intra-aortic balloon pumping after open heart surgery. ASAIO J. 1992 Jul-Sep;38(3):M574-6. doi: 10.1097/00002480-199207000-00100. PMID 1457924
- [Background] Ficek SJ, Stammers A, Deligonul U, Shurmur SW, Alonso A, Galbraith T. Hemostatic assessment of patients undergoing intraaortic balloon pump therapy. J Extra Corpor Technol. 1997 Jun;29(2):78-82. PMID 10168534
- [Background] Busch T, Sirbu H, Zenker D, Dalichau H. Vascular complications related to intraaortic balloon counterpulsation: an analysis of ten years experience. Thorac Cardiovasc Surg. 1997 Apr;45(2):55-9. doi: 10.1055/s-2007-1013687. PMID 9175219
- [Background] Todd GJ, Bregman D, Voorhees AB, Reemtsma K. Vascular complications associated with percutaneous intra-aortic balloon pumping. Arch Surg. 1983 Aug;118(8):963-4. doi: 10.1001/archsurg.1983.01390080065016. PMID 6870526
- [Background] Jiang CY, Zhao LL, Wang JA, Mohammod B. Anticoagulation therapy in intra-aortic balloon counterpulsation: does IABP really need anti-coagulation? J Zhejiang Univ Sci. 2003 Sep-Oct;4(5):607-11. doi: 10.1631/jzus.2003.0607. PMID 12958723
- [Background] Sato K, Tokairin H, Kato M. [Two patients treated with intra-aortic balloon pump counterpulsation after subarachnoid hemorrhage]. Masui. 2001 Aug;50(8):859-62. Japanese. PMID 11554017
- [Background] Vonderheide RH, Thadhani R, Kuter DJ. Association of thrombocytopenia with the use of intra-aortic balloon pumps. Am J Med. 1998 Jul;105(1):27-32. doi: 10.1016/s0002-9343(98)00128-4. PMID 9688018
- [Background] Schreiber TL, Kodali UR, O'Neill WW, Gangadharan V, Puchrowicz-Ochocki SB, Grines CL. Comparison of acute results of prophylactic intraaortic balloon pumping with cardiopulmonary support for percutaneous transluminal coronary angioplasty (PCTA). Cathet Cardiovasc Diagn. 1998 Oct;45(2):115-9. doi: 10.1002/(sici)1097-0304(199810)45:23.0.co;2-f. PMID 9786386

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intra-Aortic Balloon Pump With Heparin | Intra-Aortic Balloon Pump Without Heparin
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intra-Aortic Balloon Pump With Heparin | Intra-Aortic Balloon Pump Without Heparin | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants] — Population: Only 8 patients analyzed in Heparin group and 9 patients in non-Heparin group; data not available for remaining patients.
  Participants
    number analyzed (Participants) | 8 | 9 | 17
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 1 | 3 | 4
    >=65 years | 7 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only 8 patients analyzed in Heparin group and 9 patients in non-Heparin group; data not available for remaining patients
  Participants
    number analyzed (Participants) | 8 | 9 | 17
    Female | 1 | 4 | 5
    Male | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Minor Ischemia (Decreased Blood Flow) During the Index Hospitalization
Description: Count of participants with decreased arterial flow in lower extremity as presented by diminished pulse that resolves with balloon removal, and not resulting in any impairment of body function
Time Frame: 0-4 days post surgery
Population: Only 8 patients analyzed in Heparin group and 9 patients in non-Heparin group; data not available for remaining patients
Measure: Count of Participants; unit: Participants
Arm/Group | Intra-Aortic Balloon Pump With Heparin | Intra-Aortic Balloon Pump Without Heparin
Number analyzed (Participants) | 8 | 9
Participants | 0 | 0

2. Primary Outcome: Major Ischemia (Decreased Blood Flow) During the Index Hospitalization
Description: Count of participants with loss of Doppler signal or sensation or abnormal skin temperature, mottling or pallor in lower extremity requiring surgical intervention; or other major ischemic events including ischemic stroke; recurrent unstable ischemia (unstable angina, recurrent chest pain prompting definitive treatment such as re-percutaneous transluminal coronary angiography (PTCA), coronary artery bypass grafting (CABG), administration of thrombolytics); reinfarction including clinical symptoms or new ECG changes with creatine kinase (CK) elevation and positive creatine kinase-MB isoenzyme fraction; arterial thrombosis, embolus, dissection, or perforation; compartment syndrome; renal ischemia including new renal failure or need for dialysis; small bowel or splenic infarction; mesenteric or hepatic ischemia, or deep vein thrombosis.
Time Frame: 0-4 days post surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intra-Aortic Balloon Pump With Heparin | Intra-Aortic Balloon Pump Without Heparin
Number analyzed (Participants) | 8 | 9
Participants | 0 | 0

3. Primary Outcome: Major Bleeding During the Index Hospitalization
Description: Count of participants with hemorrhage associated with at least one of the following features as defined by the Thrombolysis in Myocardial Infarction (TIMI) Study Group criteria: Bleeding that results in a decrease in hemoglobin >/= 5g.dL or a hematocrit decrease of >/= 15% of baseline value; bleeding that is intracranial (confirmed by MRI or CT); bleeding that results in death.
Time Frame: 0-4 days post surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intra-Aortic Balloon Pump With Heparin | Intra-Aortic Balloon Pump Without Heparin
Number analyzed (Participants) | 8 | 9
Participants | 0 | 0

4. Secondary Outcome: Intra-aortic Balloon Pump-related Death During the Index Hospitalization
Time Frame: 0-4 days post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intra-Aortic Balloon Pump With Heparin | Intra-Aortic Balloon Pump Without Heparin
Number analyzed (Participants) | 23 | 23
Participants | 0 | 0

5. Secondary Outcome: Hospital Death During the Index Hospitalization
Time Frame: 0-4 post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intra-Aortic Balloon Pump With Heparin | Intra-Aortic Balloon Pump Without Heparin
Number analyzed (Participants) | 23 | 23
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Time IntraAortic Balloon Pump (IABP) was inserted in the catheterization laboratory to length of stay in hospital.. 0-4 days
Arm/Group | Intra-Aortic Balloon Pump With Heparin | Intra-Aortic Balloon Pump Without Heparin
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No